CLINICAL TRIAL: NCT02289417
Title: A Phase 2, Randomized, Placebo-controlled, Multicenter Study to Investigate the Efficacy and Safety of Apremilast (CC-10004) for Treatment of Subjects With Active Ulcerative Colitis
Brief Title: Efficacy and Safety Study of Apremilast to Treat Active Ulcerative Colitis
Acronym: UC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-UC-001; 2014-002981-64 (EudraCT Number)
Expanded Access: NCT03740516 (No longer available)
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Apremilast 30 mg PO BID (Experimental): Apremilast 30 mg by mouth (PO) twice a day (BID) for 12 weeks
  After 12 weeks:
  * Participants who achieve at least a 20% decrease from baseline in the total Mayo score (TMS) will continue to receive apremilast 30 mg BID for an additional 40 weeks. (Wk 52)
  * Participants who do not achieve at least a 20% decrease from baseline in the TMS will receive apremilast 40 mg BID for an additional 40 weeks (Wk 52)
  After 52 weeks, participants who are eligible for the Extension Phase will continue to receive the same dose of apremilast assigned at Wk 12 (30 mg BID or 40 mg BID) for an additional 52 weeks (Wk 104)
  Interventions: Drug: Apremilast
- Apremilast 40 mg PO BID (Experimental): Apremilast 40 mg by mouth (PO) twice a day (BID) for 12 weeks
  After 12 weeks, participants assigned to the 40 mg BID dose of apremilast at baseline will continue to receive apremilast 40 mg BID for an additional 40 weeks (Wk 52)
  After 52 weeks, participants who are eligible for the extension Phase will continue to receive apremilast 40 mg BID for an additional 52 weeks (Wk 104)
  Interventions: Drug: Apremilast
- Placebo BID (Placebo Comparator): Identically matching placebo by mouth (PO) twice a day (BID) for 12 weeks. After 12 weeks all participants randomized to placebo at baseline will be re-randomized to receive apremilast 30 mg or 40 mg BID for an additional 40 weeks (Wk 52)
  After Wk 52, participants who are eligible for the extension phase will continue to receive the same dose of apremilast assigned at Wk 12 (30 mg BID or 40 mg BID) for an additional 52 weeks (Wk 104)
  Interventions: Drug: Apremilast; Drug: Placebo

INTERVENTIONS:
Drug: Apremilast
  Other Names: CC-10004; Otezla
Drug: Placebo
  Arms: Placebo BID

SUMMARY:
The purpose of the study is to evaluate the clinical efficacy, safety and tolerability of apremilast (30 mg twice daily [BID] and 40 mg BID), compared with placebo, in participants with active Ulcerative Colitis (UC).

DETAILED DESCRIPTION:
Approximately 165 participants (55 subjects per arm) will be randomized in a 1:1:1 ratio to receive oral apremilast (30 mg BID or 40 mg BID), or identically appearing placebo BID for up to 12 weeks, followed by 40 weeks of blinded treatment with apremilast (30 mg BID or 40 mg BID).

At the end of the Blinded Active-treatment Phase (Week 52), participants who have a Mayo endoscopy score ≤ 1 will have the opportunity to participate in the Extension Phase. Participants enrolled in the Extension Phase will receive apremilast for an additional 52 weeks (Weeks 52 to 104). With the implementation of Amendment 4, participants entering the Extension Phase will receive apremilast 30 mg BID. Subjects currently in the Extension Phase who are receiving apremilast 40 mg BID will be switched to 30 mg BID at the next scheduled visit.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

* Male or female aged 18 and over at the time of signing the informed consent.
* Must understand and voluntarily sign an informed consent form prior to any study related assessments/procedures being conducted.
* Diagnosis of ulcerative colitis (UC) with a duration of at least 3 months prior to the Screening Visit..
* Total Mayo Score (TMS) ≥ 6 to ≤ 11 (range: 0-12) at baseline, prior to randomization in the study.
* Endoscopic subscore ≥ 2 (range: 0-3) on the Mayo score prior to randomization in the study.
* Subjects must have had a therapeutic failure, been intolerant to, or have a contraindication to, at least one of the following: oral aminosalicylates (ie, 5-aminosalicylic acid [5-ASA] compounds or sulfasalazine [SSZ]), budesonide, systemic corticosteroids, or immunosuppressants (eg, 6-mercaptopurine [6-MP], azathioprine [AZA], or methotrexate [MTX]).

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

* Diagnosis of Crohn's disease, indeterminate colitis, ischemic colitis, microscopic colitis, radiation colitis or diverticular disease-associated colitis.
* Ulcerative colitis restricted to the distal 15 cm or less (eg, ulcerative proctitis).
* Subjects who have had surgery as a treatment for UC or who, in the opinion of the Investigator, are likely to require surgery for UC during the study.
* Clinical signs suggestive of fulminant colitis or toxic megacolon.
* Prior use of any tumor necrosing factor (TNF) inhibitor (or any biologic agent).
* Prior use of mycophenolic acid, tacrolimus, sirolimus, cyclosporine or thalidomide.
* Use of intravenous (IV) corticosteroids within 2 weeks of the Screening Visit.
* Use of immunosuppressants (AZA, 6-MP or MTX) within 8 weeks of the Screening Visit.
* Use of topical treatment with 5-ASA or corticosteroid enemas or suppositories within 2 weeks of the Screening Visit.
* History of any clinically significant neurological, renal, hepatic, gastrointestinal, pulmonary, metabolic, cardiovascular, psychiatric, endocrine, hematological disorder or disease, or any other medical condition that, in the investigator's opinion, would preclude participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2019-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (99):
- United States (25):
  - Digestive Health Specialists of The Southeast, Dothan, Alabama
  - Southern California Research Institute Medical Group, Inc., Los Angeles, California
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Consultants for Clinical Research of South Florida, Boynton Beach, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Precision Clinical Research, LLC, Lauderdale Lakes, Florida
  - Pharmax Research Clinic, Inc., Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - UMass Medical Center, Worcester, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Center for Digestive Health Research, Troy, Michigan
  - Gastrointestinal Associates PA, Flowood, Mississippi
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Quality Medical Research, Nashville, Tennessee
  - Digestive Research Center/ Gastroenterology Consultants of San Antonio, Live Oak, Texas
  - Digestive Health Specialist of Tyler, Pasadena, Texas
  - San Antonio Gastroenterology, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Australia (5):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Mater Adult Hospital, South Brisbane, Queensland
  - Footscray Hospital, Footscray, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Bulgaria (7):
  - Multiprofile Hospital for Active Treatment Kaspela, Plovdiv
  - Medical Center Asklepion - Humane Medicine Research EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment ACIBADEM City Clinic Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment Sveti Ivan Rilski EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna ISUL EAD, Sofia
  - Clinic of Gastroenterology, Sofia
  - Multiprofile Hospital for Active Treatment Sveta Marina EAD, Varna
- Canada (2):
  - Winnipeg Regional Health Authority - Health Sciences Centre, Winnipeg, Manitoba
  - Hamilton Health Sciences Corporation, McMaster University Medical Centre, Hamilton, Ontario
- Czechia (4):
  - Fakultni nemocnice u sv Anny v Brne, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Hepato-Gastroenterologie HK, s. r. o., Hradec Králové
  - Nemocnice Slany, Slaný
- France (7):
  - Amiens University Hospital, Amiens
  - Hopital Beaujon, Clichy
  - CHRU Nantes, Nantes
  - CHU de Nice Archet I, Nice
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Priest-en-Jarez
  - CHRU Nancy, Vandœuvre-lès-Nancy
- Germany (4):
  - DRK Kliniken Berlin Westend, Berlin
  - Crohn-Colitis-Centre Rhein-Main, Frankfurt
  - Universitatsklinikum Schleswig-Holstein, Keil
  - Gastroenterologische Praxis Minden, Minden
- Hungary (7):
  - Pannónia Magánorvosi Centrum Kft., Budapest
  - ENDOMEDIX Kft., Budapest
  - Vasútegészségügyi Nonprofit Kiemelten Közhasznú Kft. Debreceni Egészségügyi Központja, Debrecen
  - Karolina Korhaz Rendelointezet, Mosonmagyaróvár
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Javorszky Odon Korhaz, Vác
- Italy (5):
  - Azienda Ospedaliero Universitaria Di Bologna Policlinico Sorsola Malpighi, Bologna
  - IRCCS - Istituo Clinico Humanitas - Humanitas Cancer Center, Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - Fondazione PTV Policlinico Tor Vergata, Roma
  - Complesso Integrato Columbus, Roma
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Ikazia Ziekenhuis, Rotterdam
- New Zealand (4):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato hospital, Hamilton
- Poland (11):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Osrodek Badan Klinicznych CLINSANTE S.C., Bydgoszcz
  - Centrum Medyczne sw. Lukasza, Częstochowa
  - Economicus - NZOZ ALL-MEDICUS, Katowice
  - Endoskopia Sp. z o.o., Sopot
  - Sonomed Sp. z o.o., Szczecin
  - Gastromed Kopon Zmudzinski i Wspolnicy Sp. j. Specjalistyczne Centrum Gastrologii i Endoskopii Spec. Gabinety Lekarskie, Torun
  - Centrum Zdrowia Matki, Dziecka i Mlodziezy, Warsaw
  - Niepubliczny Zaklad Opieki Zdrowotnej VIVAMED, Warsaw
  - Lexmedica Drubajlo Hanna, Wroclaw
  - Ars Medica, Wroclaw
- Russia (5):
  - Republican Clinical Hospital, Kazan'
  - Stolitsa-Medikl, LLC, Moscow
  - SEIHPE Rostov State Medical University of MoH of RF, Rostov-on-Don
  - Russian Medical Military Academy na SMKirov, Saint Petersburg
  - Regional Clinical Hospital, Saratov
- Ukraine (11):
  - Regional Clinical Hospital, Gastroenterology department, State Higher Education Institute Ivano-Frankivsk National Medical University, Ivano-Frankivsk
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Ivano-Frankivsk Central City Clinical Hospital, Ivano-Frankivsk
  - Kharkiv City Clinical Hospital 2, Kharkiv
  - Private Enterprise Private Manufacture Company Acinus, Kirovograd
  - Kremenchuk City Hospital # 1 n.a O.T.Bohaievskyi, Kremenchuk
  - Lviv Emergency Clinical Hospital, Therapeutics Department No. 1, Lviv
  - Municipal Institution Odesa Regional Clinical Hospital, Odesa
  - Central City Clinical Hospital, Uzhhorod
  - Vinnytsia Regional Clinical Hospital n a M I Pyrohov, Vinnytsia
  - Municipal Institution Zaporizhzhia, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Danese S, Neurath MF, Kopon A, Zakko SF, Simmons TC, Fogel R, Siegel CA, Panaccione R, Zhan X, Usiskin K, Chitkara D. Effects of Apremilast, an Oral Inhibitor of Phosphodiesterase 4, in a Randomized Trial of Patients With Active Ulcerative Colitis. Clin Gastroenterol Hepatol. 2020 Oct;18(11):2526-2534.e9. doi: 10.1016/j.cgh.2019.12.032. Epub 2020 Jan 8. PMID 31926340

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 61 sites in Australia (3 sites) and New Zealand (1 site); Bulgaria (6 sites), Czech Republic (2 sites), Hungary (3 sites), Poland (9 sites), Russia (1 site), and Ukraine (10 sites); Canada (2 sites) and United States (13 sites); and France (4 sites), Germany (1 site), Italy (4 sites), and the Netherlands (2 sites).
Pre-assignment Details: A total of 170 participants were randomized in a 1:1:1 ratio and received apremilast (30 mg BID or 40 mg BID), or identically appearing placebo and stratified based on concomitant use of oral corticosteroids and previous exposure to immunosuppressants.
Groups:
- Placebo: Participants were randomized to identically matching placebo capsules and received placebo capsules by mouth (PO) twice a day (BID) for 12 weeks during the double-blind placebo-controlled phase.
- Apremilast 30 mg: Participants were randomized to apremilast 30 mg capsules PO BID for 12 weeks during the double-blind placebo-controlled phase.
  At week 12, participants who achieved at least a 20% decrease from baseline in the total Mayo score (TMS) continued to receive 30 mg apremilast capsules BID for an additional 40 weeks during the active treatment phase.
- Apremilast 40 mg: Participants were randomized to 40 mg apremilast capsules PO BID for 12 weeks during the double-blind placebo-controlled phase. At week 12, participants who achieved at least a 20% decrease from baseline in the TMS continued to receive 40 mg apremilast capsules BID for an additional 40 weeks during the active treatment phase.
- Placebo/Apremilast 30 mg: Participants initially randomized to placebo capsules in the placebo-controlled period were re-randomized at week 12 to receive 30 mg apremilast capsules BID for 40 weeks during the active treatment phase.
- Placebo/Apremilast 40 mg: Participants initially randomized to placebo in the placebo-controlled period were re-randomized at week 12 to receive 40 mg apremilast capsules BID for 40 weeks during the active treatment phase.
- Apremilast 30 mg/Apremilast 40 mg: Participants initially randomized to 30 mg apremilast capsules BID in the placebo-controlled phase who did not achieve at least a 20% decrease from baseline in the TMS were re-assigned to 40 mg apremilast capsules BID for 40 weeks during the active treatment phase.
- Apremilast 40 mg/ Apremilast 40 mg: Participants initially randomized to 40 mg apremilast capsules BID in the placebo-controlled phase who did not achieve at least a 20% decrease from baseline in the TMS continued to receive 40 mg apremilast capsules BID for an additional 40 weeks during the active treatment phase.
- Extension Phase: Apremilast 30 mg: Participants who completed 52 weeks of treatment and had a Mayo endoscopy score ≤ 1 at week 52 were eligible to participate in the 52-week extension phase and receive 30 mg apremilast BID for an additional 52 weeks. This includes participants assigned to 30 mg apremilast BID at week 12, and participants who entered the extension phase after implementation of Protocol Amendment 4.
- Extension Phase Apremilast 40 mg: Participants who completed 52 weeks of treatment and had a Mayo endoscopy score ≤ 1 at week 52 were eligible to participate in the 52-week extension phase and receive 40 mg apremilast BID for an additional 52 weeks. After implementation of Protocol Amendment 4 participants were switched to 30 mg apremilast BID for the remainder of the extension phase.
Period: Placebo-Controlled Phase Weeks 0-12
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg | Placebo/Apremilast 30 mg | Placebo/Apremilast 40 mg | Apremilast 30 mg/Apremilast 40 mg | Apremilast 40 mg/ Apremilast 40 mg | Extension Phase: Apremilast 30 mg | Extension Phase Apremilast 40 mg
Started | 58 | 57 | 55 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 51 | 53 | 52 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Active Treatment Phase Weeks 12-52
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg | Placebo/Apremilast 30 mg | Placebo/Apremilast 40 mg | Apremilast 30 mg/Apremilast 40 mg | Apremilast 40 mg/ Apremilast 40 mg | Extension Phase: Apremilast 30 mg | Extension Phase Apremilast 40 mg
Started | 0 | 41 | 42 | 26 | 25 | 12 (1 participant went only to Week 20) | 7 (Week 12 TMS were missing for 3 participants) | 0 | 0
Completed | 0 | 39 | 32 | 17 | 20 | 7 | 5 | 0 | 0
Not Completed | 0 | 2 | 10 | 9 | 5 | 5 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 4 | 2 | 2 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 4 | 6 | 2 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Period: Extension Phase Weeks 52-104
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg | Placebo/Apremilast 30 mg | Placebo/Apremilast 40 mg | Apremilast 30 mg/Apremilast 40 mg | Apremilast 40 mg/ Apremilast 40 mg | Extension Phase: Apremilast 30 mg | Extension Phase Apremilast 40 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 45 | 54
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 38 | 48
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population consisted of all participants who were randomized and received at least 1 dose of investigational product (IP).
Groups:
- Placebo: Participants were randomized to identically matching placebo capsules and received placebo capsules by mouth PO BID for 12 weeks during the double-blind placebo-controlled phase.
- Apremilast 30 mg: Participants were randomized to apremilast 30 mg capsules PO BID for 12 weeks during the double-blind placebo-controlled phase.
- Apremilast 40 mg: Participants were randomized to 40 mg apremilast capsules PO BID for 12 weeks during the double-blind placebo-controlled phase.
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg | Total
Number analyzed (Participants) | 58 | 57 | 55 | 170
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.9 (14.04) | 40.1 (13.50) | 43.4 (14.92) | 42.1 (14.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 21 | 64
  Male | 33 | 39 | 34 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 5 | 8
  Not Hispanic or Latino | 55 | 54 | 46 | 155
  Unknown or Not Reported | 1 | 2 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 1
  White | 54 | 52 | 45 | 151
  Other | 1 | 1 | 1 | 3
  Not Reported or Collected | 3 | 4 | 8 | 15
Duration of Ulcerative Colitis [Mean (Standard Deviation); unit: Years] | 6.85 (7.043) | 6.15 (5.432) | 8.63 (10.278) | 7.19 (7.832)
Baseline Total Mayo Score (TMS) [Mean (Standard Deviation); unit: units on a scale] — The TMS is an instrument designed to measure disease activity of Ulcerative Colitis (UC). The Mayo score ranges from 0 to 12 points. It consists of 4 subscores, each graded from 0 to 3 with higher scores indicating more severe disease:
  * Stool Frequency Subscore (SFS)
  * Rectal Bleeding Subscore (RBS)
  * Endoscopy Subscore
  * Physician's Global Assessment (PGA)
  units on a scale | 8.2 (1.68) | 8.5 (1.62) | 8.1 (1.67) | 8.3 (1.65)
Modified Mayo Score (MMS) [Mean (Standard Deviation); unit: units on a scale] — The MMS was based on the stool frequency, rectal bleeding and endoscopy subscores of the total Mayo score, and excluded the Physician's Global subscore, since this was a global measure that is subjective in nature. The MMS range from 0 to 9 points with zero indicating no symptoms of active ulcerative colitis and 9 indicating the most severe symptoms.
  units on a scale | 6.1 (1.51) | 6.4 (1.48) | 6.0 (1.47) | 6.2 (1.49)
Partial Mayo Score (PMS) [Mean (Standard Deviation); unit: units on a scale] — The partial Mayo score is the sum of the rectal bleeding score, the stool frequency score and the physician's global assessment. The partial Mayo score range is from 0 to 9 points with zero indicating no symptoms of active ulcerative colitis and 9 indicating the most severe symptoms and assessment.
  units on a scale | 5.6 (1.46) | 5.8 (1.44) | 5.5 (1.57) | 5.6 (1.49)
Mayo Endoscopic Subscore (MES) [Mean (Standard Deviation); unit: units on a scale] — The Mayo endoscopy subscore findings are defined as:
  0 = Normal or inactive disease
  1. = Mild Disease (erythema, decreased vascular pattern, mild friability)
  2. = Moderate Disease (marked erythema, lack of vascular pattern, friability erosions) 3 = Severe Disease (spontaneous bleeding, ulceration).
  units on a scale | 2.6 (0.49) | 2.7 (0.45) | 2.6 (0.49) | 2.6 (0.48)
Baseline Use of Oral Corticosteroids [Number; unit: Participants] — Participants were stratified based on concomitant use of oral corticosteroids and previous exposure to immunosuppressants.
  Participants | 17 | 14 | 12 | 43
Previous Exposure to Use of Immunosuppressants [Number; unit: Participants] — Participants were stratified based on concomitant use of oral corticosteroids and previous exposure to immunosuppressants.
  Participants | 17 | 18 | 16 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Clinical Remission by Total Mayo Score (TMS) at Week 12
Description: Clinical remission was defined as a total Mayo score ≤ 2 points, with no individual subscore exceeding 1 point. The TMS is an instrument designed to measure disease activity of UC. The Mayo score ranges from 0 to 12 points. It consists of 4 subscores, each graded from 0 to 3 with higher scores indicating more severe disease.
  * Stool Frequency Subscore (SFS)
  * Rectal Bleeding Subscore (RBS)
  * Endoscopy Subscore
  * Physician's Global Assessment (PGA). Two-sided 95% confidence intervals (CI) for the within-group percentages are based on the Wilson score method.
Time Frame: Week 12
Population: The intent to treat (ITT) population included all participants who received at least one dose of IP. Participants with insufficient data for response determination were considered non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 58 | 57 | 55
Percentage of Participants | 12.1 [6.0 to 22.9] | 31.6 [21.0 to 44.5] | 21.8 [12.9 to 34.4]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0142, Cochran-Mantel-Haenszel; Stratification was based on baseline use of oral (PO) corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 19.2, 95% CI 2-sided [3.4 to 33.6] — Stratified difference in percentages is the weighted average of the treatment differences across the strata with the CMH weights, with 2-sided 95% CI based on the stratified Newcombe method
Statistical Analysis 2: Comparison: Placebo vs Apremilast 40 mg; Test type: Superiority; p = 0.2689, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 7.7, 95% CI 2-sided [-6.9 to 22.0] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants Who Achieved a Clinical Response by Total Mayo Score and the Reduction in the Rectal Bleeding Subscore at Week 12
Description: Clinical response was defined as a decrease from baseline in the TMS of at least 3 points and at least 30%, along with a reduction in the rectal bleeding subscore (RBS) of at least 1 point or an absolute RBS of ≤ 1. The TMS is an instrument designed to measure disease activity of UC. The Mayo score ranges from 0 to 12 points. It consists of 4 subscores, each graded from 0 to 3 with higher scores indicating more severe disease.
  * Stool Frequency Subscore (SFS)
  * Rectal Bleeding Subscore
  * Endoscopy Subscore
  * Physician's Global Assessment (PGA)
  Rectal bleeding (subscore 0-3) was defined as:
  0 = No blood seen
  1. = Streaks of blood with stool less than half the time
  2. = Obvious blood with stool
  3. = Blood alone passes Two-sided 95% CI for the within-group percentages are based on the Wilson score method.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 58 | 57 | 55
Percentage of Participants | 46.6 [34.3 to 59.2] | 61.4 [48.4 to 72.9] | 67.3 [54.1 to 78.2]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.1224, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 14.6, 95% CI 2-sided [-3.6 to 31.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 40 mg; Test type: Superiority; p = 0.0401, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 19.4, 95% CI 2-sided [1.1 to 36.0] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Who Achieved an Endoscopic Remission at Week 12
Description: An endoscopic remission was defined as a Mayo endoscopic subscore (MES) of 0 at Week 12.
  The MES subscore findings were defined as:
  0 = Normal or inactive disease
  1. = Mild Disease (erythema, decreased vascular pattern, mild friability)
  2. = Moderate Disease (marked erythema, lack of vascular pattern, friability erosions)
  3. = Severe Disease (spontaneous bleeding, ulceration)
  The endoscopy subscores consisted of findings that were centrally read through proctosigmoidoscopy, graded from 0 to 3 with higher scores indicating more severe disease. Two-sided 95% CIs for the within-group percentage were based on the Wilson score method.
Time Frame: Week 12
Population: The intent to treat population included all participants who received at least one dose of IP. Participants with insufficient data for response determination were considered non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 58 | 57 | 55
Percentage of Participants | 3.4 [1.0 to 11.7] | 8.8 [3.8 to 18.9] | 7.3 [2.9 to 17.3]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.2472, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 5.2, 95% CI 2-sided [-5.7 to 16.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 40 mg; Test type: Superiority; p = 0.4628, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 3.1, 95% CI 2-sided [-7.5 to 14.6] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants Who Achieved an Endoscopic Response at Week 12
Description: An endoscopic response is defined as a decrease from baseline of at least 1 point in the MES at Week 12. The Mayo endoscopy subscore findings were defined as:
  0 = Normal or inactive disease
  1. = Mild Disease (erythema, decreased vascular pattern, mild friability)
  2. = Moderate Disease (marked erythema, lack of vascular pattern, friability erosions) 3 = Severe Disease (spontaneous bleeding, ulceration).
  The endoscopy subscores consisted of findings that were centrally read through proctosigmoidoscopy, graded from 0 to 3 with higher scores indicating more severe disease. Two-sided 95% CIs for the within-group percentage were based on the Wilson score method.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 58 | 57 | 55
Percentage of Participants | 41.4 [29.6 to 54.2] | 73.7 [61.0 to 83.4] | 47.3 [34.7 to 60.2]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 32.0, 95% CI 2-sided [13.8 to 47.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 40 mg; Test type: Superiority; p = 0.6878, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 3.7, 95% CI 2-sided [-14.4 to 21.5] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants Who Achieved a Rectal Bleeding Subscore (RBS) of ≤ 1 at Week 12
Description: The RBS was measured as:
  0 = No blood seen
  1. = Streaks of blood with stool less than half the time
  2. = Obvious blood with stool most of the time
  3. = Blood alone passes
  The daily bleeding score represents the most severe bleeding of the day. Two-sided 95% CI for the within-group proportions are based on the Wilson score method.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 58 | 57 | 55
Percentage of Participants | 72.4 [59.8 to 82.2] | 84.2 [72.6 to 91.5] | 87.3 [76.0 to 93.7]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.1388, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 11.5, 95% CI 2-sided [-4.1 to 26.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 40 mg; Test type: Superiority; p = 0.0788, Cochran-Mantel-Haenszel — Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 13.5, 95% CI 2-sided [-1.6 to 27.7] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission in the Modified Mayo Subscore (MMS) at Week 12
Description: Clinical remission was defined as a modified Mayo score of ≤ 2, with no individual subscore > 1, at Week 12. The MMS was based on a modification of the total Mayo score (TMS) which included the stool frequency, rectal bleeding, and endoscopic subscores of the TMS and excluded the Physician's Global Assessment (PGA) subscore, since this was a global measure that is subjective in nature. The MMS ranges from 0 to 9 points with higher scores indicating greater disease severity. The endoscopy subscores was centrally reviewed. Two-sided confidence intervals for the within-group percentage were based on the Wilson score method.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 58 | 57 | 55
Percentage of Participants | 19.0 [10.9 to 30.9] | 43.9 [31.8 to 56.7] | 27.3 [17.3 to 40.2]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0046, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 24.8, 95% CI 2-sided [7.5 to 40.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 40 mg; Test type: Superiority; p = 0.4476, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 6.0, 95% CI [-9.8 to 21.6] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response in the Modified Mayo Subscore (MMS) at Week 12
Description: Clinical response in the MMS was defined as a decrease from baseline in the MMS of at least 2 points and at least 25%, along with a reduction in the RBS of at least 1 point or an absolute RBS ≤ 1. The MMS was based on the stool frequency, rectal bleeding, and endoscopic subscores of the TMS and excluded the PGA subscore. The MMS ranges from 0 to 9 points with higher scores indicating greater disease severity.
  The RBS was measured as:
  0 = No blood seen
  1. = Streaks of blood with stool less than half the time
  2. = Obvious blood with stool most of the time
  3. = Blood alone passes
  The daily bleeding score represents the most severe bleeding of the day. The endoscopy subscores was centrally reviewed. Two-sided confidence intervals for the within-group percentage were based on the Wilson score method.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 58 | 57 | 55
Percentage of Participants | 46.6 [34.3 to 59.2] | 63.2 [50.2 to 74.5] | 67.3 [54.1 to 78.2]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0755, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 16.7, 95% CI 2-sided [-1.4 to 33.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 40 mg; Test type: Superiority; p = 0.0370, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 19.8, 95% CI 2-sided [1.5 to 36.4] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission in the Partial Mayo Subscore (PMS) With no Individual Subscore >1 at Week 8
Description: Clinical remission in the partial Mayo subscore was defined as a PMS of 2 points or lower, with no individual subscore >1. The PMS is a discrete ordinal scale ranging from 0 (normal or inactive disease) to 9 (severe disease) and is a composite of 3 subscores:
  Stool Frequency Subscore, Rectal Bleeding Subscore, and Physician's Global Assessment Subscore, each of which ranges from 0 (normal) to 3 (severe disease).
  Two-sided 95% CI for the within-group proportions are based on the Wilson score method.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 58 | 57 | 55
Percentage of Participants | 32.8 [22.1 to 45.6] | 47.4 [35.0 to 60.1] | 52.7 [39.8 to 65.3]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.1167, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 14.6, 95% CI 2-sided [-3.3 to 31.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 40 mg; Test type: Superiority; p = 0.0534, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 18.1, 95% CI 2-sided [-0.3 to 34.9] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response in the Partial Mayo Subscore at Week 8
Description: Clinical response in the PMS was defined as a decrease from baseline in PMS of at least 2 points and at least 25%, with an accompanying decrease in the RBS of at least 1 point or an absolute RBS of 0 or 1. The PMS score is a discrete ordinal scale ranging from 0 (normal or inactive disease) to 9 (severe disease) and is a composite of 3 subscores:
  Stool Frequency Subscore, Rectal Bleeding Subscore, and Physician's Global Assessment Subscore, each of which ranges from 0 (normal) to 3 (severe disease).
  Two-sided 95% CI for the within-group proportions are based on the Wilson score method.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 58 | 57 | 55
Percentage of Participants | 48.3 [35.9 to 60.8] | 64.9 [51.9 to 76.0] | 81.8 [69.7 to 89.8]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0758, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 16.6, 95% CI 2-sided [-1.5 to 33.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 40 mg; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel; Stratification was based on baseline use of PO corticosteroids and previously used immunosuppressants (yes/no); Stratified Difference = 32.5, 95% CI 2-sided [14.9 to 47.5] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: The Number of Participants Who Experienced Treatment Emergent Adverse Events (TEAEs) During the Placebo-Controlled Phase
Description: A TEAE was defined as any adverse event (AE) occurring or worsening on or after the first treatment of apremilast and up to 28 days after the last apremilast dose or the last follow-up date, whichever occurred earlier. A serious AE = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. The severity of AEs was assessed by the investigator and based on the following scale: Mild = asymptomatic or mild symptoms; clinical or diagnostic observations only; Moderate = Symptoms cause moderate discomfort; Severe (could be non-serious or serious) = symptoms causing severe discomfort/pain
Time Frame: From the first dose of investigational product (IP) and no later than 28 days after the last dose of IP for those who had completed the study or discontinued (D/C) early; maximum duration of exposure to treatment was 12.00 weeks
Population: Safety population included all participants who were enrolled and received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 58 | 57 | 55
Participants
  Any TEAE | 31 | 28 | 36
  Any IP-related TEAE | 12 | 13 | 20
  Any Severe TEAE | 4 | 0 | 1
  Any Serious TEAE | 2 | 0 | 1
  Any Serious IP-related TEAE | 0 | 0 | 0
  Any TEAE Leading to IP Withdrawal | 5 | 0 | 1
  Any TEAE Leading to IP Interruption | 1 | 0 | 0
  Any TEAE Leading to Death | 0 | 0 | 0

11. Secondary Outcome: The Number of Participants Who Discontinued Apremilast Due to Treatment Emergent Adverse Events During the Placebo-Controlled Period
Description: A TEAE was defined as any AE occurring or worsening on or after the first treatment of apremilast and up to 28 days after the last apremilast dose or the last follow-up date, whichever occurred earlier. A serious AE = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. The severity of AEs was assessed by the investigator and based on the following scale: Mild = asymptomatic or mild symptoms; clinical or diagnostic observations only; Moderate = Symptoms cause moderate discomfort; Severe (could be non-serious or serious) = symptoms causing severe discomfort/pain.
Time Frame: From the first dose of IP and no later than 28 days after the last dose of IP for those who had completed the study or discontinued early; median duration of exposure to treatment was 12.00 weeks
Population: Safety population included all participants who were enrolled and received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 58 | 57 | 55
Participants | 5 | 0 | 1

12. Secondary Outcome: The Number of Participants Who Experienced TEAEs During the Apremilast (APR) Exposure Period (Active Treatment Phase) Through Week 52
Description: as for outcome 11
Time Frame: From first dose of IP and no later than 28 days after last dose of IP for those who completed the active treatment phase or D/C early; median duration of exposure = 41.00, 44.15 and 40.00 weeks respectively for 30 mg, 40 mg and 30 mg/40 mg APR arms
Population: Apremilast exposure population included all participants who were randomized at Week 0 or assigned at Week 12 to an apremilast group and received at least 1 dose of apremilast.
Measure: Count of Participants; unit: Participants
Groups:
- Apremilast 30 mg: TEAEs during the apremilast 30 mg BID treatment for participants who received 30 mg apremilast capsules BID only and participants who initially received 30 mg apremilast capsules BID and switched to 40 mg apremilast capsules BID at Week 12, and participants who initially received placebo capsules BID and switched to 30 mg apremilast capsules BID at Week 12.
- Apremilast 40 mg: TEAEs during the apremilast 40 mg BID treatment for participants who received 40 mg apremilast capsules BID only, and participants who initially received placebo BID and switched to 40 mg apremilast capsules BID at Week 12.
- Apremilast 30 mg/Apremilast 40 mg: TEAEs during the apremilast 40 mg BID treatment for participants who initially received 30 mg apremilast BID and switched to apremilast 40 mg BID at Week 12.
Arm/Group | Apremilast 30 mg | Apremilast 40 mg | Apremilast 30 mg/Apremilast 40 mg
Number analyzed (Participants) | 83 | 80 | 11
Participants
  Any TEAE | 60 | 67 | 8
  Any Severe TEAE | 5 | 6 | 0
  Any Serious TEAE | 6 | 8 | 1
  Any TEAE Leading to Drug Withdrawal | 3 | 9 | 1
  Any TEAE Leading to Drug Interruption | 1 | 4 | 0
  Any TEAE Leading to Death | 0 | 0 | 0

13. Secondary Outcome: The Number of Participants Who Experienced TEAEs During Week 52 to Week 104 (Extension Phase)
Description: as for outcome 11
Time Frame: From the first dose of IP at Week 52 and no later than 28 days after the last dose of IP for those who completed the study or had discontinued early; median exposure of apremilast for the total apremilast group was 52 weeks.
Population: Participants who received at least 1 dose of apremilast after week 52.
Measure: Count of Participants; unit: Participants
Groups:
- Extension Phase: Apremilast 30 mg: Participants who completed 52 weeks of treatment and had a Mayo endoscopy score ≤ 1 at week 52 were eligible to participate in the 52-week extension phase and received 30 mg apremilast BID for an additional 52 weeks. Includes participants assigned to 30 mg apremilast BID at week 12, and participants who entered the extension phase after implementation of Protocol Amendment 4.
- Extension Phase: Apremilast 40 mg: Participants who completed 52 weeks of treatment and had a Mayo endoscopy score ≤ 1 at week 52 were eligible to participate in the 52-week extension phase and received 40 mg apremilast BID for an additional 52 weeks. After implementation of Protocol Amendment 4, participants were switched to 30 mg apremilast BID for the remainder of the extension phase.
Arm/Group | Extension Phase: Apremilast 30 mg | Extension Phase: Apremilast 40 mg
Number analyzed (Participants) | 45 | 54
Participants
  Any TEAE | 16 | 27
  Any Severe TEAE | 1 | 0
  Any Serious TEAE | 4 | 3
  Any Serious IP-related TEAE | 0 | 1
  Any TEAE Leading to IP Withdrawal | 2 | 1
  Any TEAE Leading to IP Interruption | 1 | 0
  Any TEAE Leading to Death | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of IP and no later than 28 days after the last dose of IP for those who had completed the study or discontinued early. AEs are reported for the placebo-controlled phase from Week 0 to Week 12 and for the apremilast exposure period from Week 0 to Week 104.
Description: Median duration of study drug was 12 weeks in the placebo controlled phase, 41.00, 44.15 and 40.00 weeks respectively for 30 mg, 40 mg and 30 mg/40 mg APR arms in the active treatment phase and 52 weeks in the extension phase. MedDRA Version 20.1 was utilized in the placebo controlled phase and Version 22 in the active treatment and extension phase.
Groups:
- Placebo (Placebo Controlled Period): TEAEs for participants who were randomized to identically matching placebo capsules twice a day (BID) for 12 weeks during the double-blind placebo-controlled phase.
- Apremilast 30 mg (Placebo Controlled Period): TEAEs for participants who were randomized to apremilast 30 mg capsules PO BID for 12 weeks during the double-blind placebo-controlled phase.
- Apremilast 40 mg BID (Placebo Controlled Period): TEAEs for participants who were randomized to apremilast 40 mg capsules PO BID for 12 weeks during the double-blind placebo-controlled phase.
- Apremilast 30 mg (Apremilast Exposure Period): TEAEs during the apremilast 30 mg BID treatment for participants who received 30 mg apremilast capsules BID only and participants who initially received 30 mg apremilast capsules BID and switched to 40 mg apremilast capsules BID at Week 12, and participants who initially received placebo capsules BID and switched to 30 mg apremilast capsules BID at Week 12.
- Apremilast 40 mg (Apremilast Exposure Period): TEAEs during the apremilast 40 mg BID treatment for participants who received 40 mg apremilast capsules BID only, and participants who initially received placebo BID and switched to 40 mg apremilast capsules BID at Week 12.
- Apremilast 30/40 mg (Apremilast Exposure Period): TEAEs during the apremilast 40 mg BID treatment for participants who initially received 30 mg apremilast BID and switched to apremilast 40 mg BID at Week 12. for participants who initially received 30 mg apremilast dosage and switched to 40 mg apremilast capsules BID at Week 12.
Arm/Group | Placebo (Placebo Controlled Period) | Apremilast 30 mg (Placebo Controlled Period) | Apremilast 40 mg BID (Placebo Controlled Period) | Apremilast 30 mg (Apremilast Exposure Period) | Apremilast 40 mg (Apremilast Exposure Period) | Apremilast 30/40 mg (Apremilast Exposure Period)
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/57 | 0/55 | 0/83 | 0/80 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/58 | 0/57 | 1/55 | 9/83 | 11/80 | 1/11
Other Adverse Events (participants affected / at risk) | 20/58 | 26/57 | 25/55 | 49/83 | 53/80 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Placebo Controlled Period) (N=58) | Apremilast 30 mg (Placebo Controlled Period) (N=57) | Apremilast 40 mg BID (Placebo Controlled Period) (N=55) | Apremilast 30 mg (Apremilast Exposure Period) (N=83) | Apremilast 40 mg (Apremilast Exposure Period) (N=80) | Apremilast 30/40 mg (Apremilast Exposure Period) (N=11)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 3 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Epididymitis tuberculous (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epididymal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Placebo Controlled Period) (N=58) | Apremilast 30 mg (Placebo Controlled Period) (N=57) | Apremilast 40 mg BID (Placebo Controlled Period) (N=55) | Apremilast 30 mg (Apremilast Exposure Period) (N=83) | Apremilast 40 mg (Apremilast Exposure Period) (N=80) | Apremilast 30/40 mg (Apremilast Exposure Period) (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 4 | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 3 | 6 | 8 | 9 | 3
Asthenia (General disorders) | 2 | 3 | 1 | 5 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 4 | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 0 | 4 | 3 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 5 | 6 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 4 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 3 | 3 | 3
Influenza like illness (General disorders) | 0 | 1 | 1 | 2 | 2 | 1
Pyrexia (General disorders) | 2 | 1 | 1 | 1 | 2 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 3 | 3 | 1
Influenza (Infections and infestations) | 1 | 0 | 1 | 2 | 3 | 1
Nasopharyngitis (Infections and infestations) | 1 | 4 | 2 | 7 | 8 | 2
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 4 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Faecal calprotectin increased (Investigations) | 0 | 1 | 1 | 1 | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 5 | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 3 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 4 | 12 | 14 | 17 | 25 | 2
Migraine (Nervous system disorders) | 0 | 1 | 1 | 2 | 3 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 2 | 4 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 1 | 3 | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 5 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1
Angiopathy (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT02289417/SAP_001.pdf
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT02289417/Prot_002.pdf